CLINICAL TRIAL: NCT01873716
Title: Indocyanine Green Fluorescence Uptake in Human Carotid Artery Plaque -- A Pilot Study
Brief Title: Indocyanine Green Fluorescence Uptake in Human Carotid Artery Plaque
Acronym: BRIGHT-CEA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Farouc Amin Jaffer, Associate Professor of Medicine, Harvard Medical School, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012P000895
Record Dates: First submitted 2013-05-23; First posted 2013-06-10 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Atherosclerosis; Atherosclerotic Plaque; Carotid Stenosis
Keywords: Atherosclerosis; Molecular Imaging; Vascular Biology; Inflammation; Fluorescence
MeSH Terms: conditions — Atherosclerosis; Plaque, Atherosclerotic; Carotid Stenosis; Inflammation | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Injection of Indocyanine Green (Experimental): Injection of Indocyanine Green prior to carotid endarterectomy surgery. Collection of specimen during surgery with subsequent carotid tissue analysis.
  Interventions: Drug: Indocyanine green
- No injection (No Intervention): No injection prior to carotid endarterectomy surgery. Collection of specimen during surgery with subsequent carotid tissue analysis.

INTERVENTIONS:
Drug: Indocyanine green — Indocyanine green (ICG) for injection, 0.25mg/kg intravenously. A maximum of 25mg is given, approximately 30-60 minutes before carotid endarterectomy
  Other Names: FDA Application No. (ANDA) 040811
  Arms: Injection of Indocyanine Green

SUMMARY:
This will be a pilot study of 9 patients undergoing standard-of-care clinically indicated carotid endarterectomy. The nine patients will receive an injection of Indocyanine green (ICG) at a dose of 0.25 mg/kg (maximum 25 mg) as an intravenous bolus.

Immediately following endarterectomy, the resected specimen will be immersed in normal saline. Ex vivo fluorescence reflectance imaging (FRI) and immunohistochemistry will be performed.

The investigators hypothesize that compared to controls, ICG-injected patients will demonstrate increased ex vivo and microscopic ICG fluorescence signal within areas of plaque.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients scheduled for elective carotid endarterectomy at Massachusetts General Hospital
* Age > 18 years of age.
* Signed informed consent.

Exclusion criteria:

* Hemodynamic instability
* Any history of iodide allergy
* Any history of renal failure (estimated Glomerular Filtration Rate (eGFR) <50 ml/min/1.73 m2)
* Any history of liver failure
* Any history of bleeding diathesis
* Any history of cerebral vascular accident in the preceding 3 months
* Pregnant or lactating females.
* Hx of seafood allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Tissue uptake of indocyanine green in carotid plaque | within 3 months after carotid endarterectomy
  Characterize tissue distribution of indocyanine green in human carotid artery specimens after carotid endarterectomy using fluorescence microcopy

SECONDARY OUTCOMES:
Relationship of indocyanine green uptake to carotid plaque histology | within 3 months after carotid endarterectomy
  Analysis of tissue distribution of indocyanine green in human carotid artery specimens after carotid endarterectomy using histopathology

CONTACTS AND LOCATIONS:
Overall Officials: Farouc A Jaffer, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Vinegoni C, Botnaru I, Aikawa E, Calfon MA, Iwamoto Y, Folco EJ, Ntziachristos V, Weissleder R, Libby P, Jaffer FA. Indocyanine green enables near-infrared fluorescence imaging of lipid-rich, inflamed atherosclerotic plaques. Sci Transl Med. 2011 May 25;3(84):84ra45. doi: 10.1126/scitranslmed.3001577. PMID 21613624
- [Derived] Verjans JW, Osborn EA, Ughi GJ, Calfon Press MA, Hamidi E, Antoniadis AP, Papafaklis MI, Conrad MF, Libby P, Stone PH, Cambria RP, Tearney GJ, Jaffer FA. Targeted Near-Infrared Fluorescence Imaging of Atherosclerosis: Clinical and Intracoronary Evaluation of Indocyanine Green. JACC Cardiovasc Imaging. 2016 Sep;9(9):1087-1095. doi: 10.1016/j.jcmg.2016.01.034. Epub 2016 Aug 17. PMID 27544892